CLINICAL TRIAL: NCT06666621
Title: Antagonism of Endogenous Opioids: Use in Interpretation of Injections
Brief Title: Endogenous Opioid Response to Injections
Acronym: AEOUI2
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Middle Tennessee Research Institute (Other)
Collaborators: International Pain and Spine Intervention Society (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1792559; Foundation Grant (Other: International Pain and Spine Intervention Society)
Record Dates: First submitted 2024-10-23; First posted 2024-10-30 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Low Back Pain; Zygapophyseal Joint Arthritis
Keywords: low back pain; zygapophysial joint arthritis; endogenous opioids; lumbar medial branch block
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: prospective, within-subject
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single arm study: endogenous opioid blockade (Other): This is a single group study. The participants will undergo two sequential experimental conditions: saline infusion and naloxone infusion.
  Participants will be identified as candidates for standard of care lumbar medial branch block, consented, and enrolled. Baseline demographics and patient reported clinical measures will be collected.
  All participants will have IV placed, undergo standard of care lumbar medial branch block, wait 20 minutes, then have their response to procedure assessed. Then normal saline will be infused through the IV over several minutes, 10 minutes will pass, and response to procedure re-assessed. Then naloxone will be infused through the IV over several minutes, 10 minutes will pass, and response to procedure re-assessed for a final time. IV will then be removed.
  Participants will then follow standard of care clinical practice for second lumbar medial branch block and lumbar medial branch radiofrequency neurotomy treatment.
  Interventions: Drug: Normal saline infusion; Drug: Naloxone infusion

INTERVENTIONS:
Drug: Normal saline infusion — After assessment of response to lumbar medial branch block, 8 ml normal saline will be infused through IV over several minutes. 10 minutes will pass, and response to lumbar medial branch block procedure will be re-assessed.
  After this step, naloxone infusion will occur (see next intervention)
Drug: Naloxone infusion — After infusion of normal saline and re-assessment of response to lumbar medial branch block procedure, 8 milligrams of naloxone will be infused over several minutes. Then after 10 minutes, response to lumbar medial branch block procedure will be re-reassessed for the final time.

SUMMARY:
This study will study pain relief after spine injections that are used to guide care. Some improvements in pain from a procedure might be from placebo effect rather than the physiological effect of the procedure. The study will use naloxone to reverse the effect of the body's internal placebo system after a spine injection, so the placebo effect and the injection effect can be measured separately. This process may improve the understanding of spine injections and their ability to guide pain care.

DETAILED DESCRIPTION:
Nerve blocks are commonly used in pain medicine to diagnose painful conditions and predict response to invasive procedures and surgeries. Placebo responses may cripple clinicians' ability to interpret responses to nerve blocks and guide patient care, when reported pain relief is due to placebo rather than the nerve block.

Existing methods to assess placebo response in clinical practice are limited and indirect. The area that is most explored is in the diagnosis of pain from the facet joints of the spine and relies on an indirect signal from repeated diagnostic injections.

Lumbar medial branch radiofrequency neurotomy (LMBRN) is commonly used to treat low back pain and can lead to large improvements in pain and disability. There is a high failure rate of LMBRN even after a series of controlled prognostic injections called lumbar medial branch nerve blocks (LMBB) with local anesthetic. The discrepancy between response to LMBB and LMBRN has been attributed to the confounding of pain relief from the nerve block with pain relief from the placebo response.

Endogenous opioids (EO), substances produced within the human body that bind to opioid receptors and produce opioid analgesia, are likely responsible for most of the placebo response caused by LMBB.

This study will use naloxone, an opioid receptor antagonist, to completely block the activity of EOs in patients. First, the pain relief after LMBB will be recorded - this is a combination of the effect of the nerve block and EO released in the placebo response. Normal saline will be infused, as an internal control for the state of receiving an infusion. Naloxone will then be infused, reversing EO-dependent placebo analgesia - the analgesia remaining will be from the nerve block. Finally, clinical outcomes from LMBRN will be collected to determine whether using naloxone with LMBB can improve prediction of outcomes with LMBRN.

Naloxone will be used to probe a mechanism of procedurally-induced endogenous-opioid mediated placebo analgesia. No IND is pursued in this study.

These data will provide detailed parameters of placebo response from LMBB, improving interpretation of LMBB for estimation of prevalence of zygapophyseal joint pain and for prognostication of LMBRN.

Furthermore, if this methodology of EO reversible analgesia is feasible for investigation of placebo from LMBB, it will be more broadly investigated in diagnostic and prognostic injections used in interventional pain management.

ELIGIBILITY:
Inclusion Criteria:

* Capable of understanding and providing consent in English and capable of complying with the outcome instruments used
* ≥3 months low back pain with persistent limiting symptoms despite conventional treatment (physical therapy and oral medications)
* Low back pain NRS ≥ 4/10 in intensity on 7-day average and at time of lumbar medial branch block

Exclusion Criteria:

* Daily use of opioid medications or recreational drugs, or if using opioids PRN, report of opioid use within the 3 days prior to participating in the protocol
* Positive urine drug screen for opioid medication on the day of naloxone administration
* Allergy to naloxone
* Refusal of or failure to place IV
* Previous LMBB or LMBRN
* Known spine condition that may affect the ability to diagnose or treat facet pain or lead to spine surgery (e.g. instability, severe spinal stenosis, radiculopathy, previous spine operation resulting in alteration of anatomy targeted by LMBB or LMBRFN)
* Active medical condition that would limit the safety of naloxone administration (e.g. severe kidney or liver failure, unstable cardiac disease, infection, severe coagulopathy)
* Psychiatric, medical, neurologic, or pain-related disorder that may compromise the ability of the patient to accurately report changes in low back pain
* Requirement for procedural sedation to tolerate LMBB

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2024-08-22 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Endogenous opioid-dependent placebo analgesia | 10 minutes after naloxone infusion
  Endogenous opioid-dependent placebo analgesia is defined as change in analgesia after lumbar medial branch block #1 (measured by numeric pain rating scale) after infusing naloxone

SECONDARY OUTCOMES:
Saline-reversible analgesia | 10 minutes after saline infusion
  Saline-reversible analgesia is defined as change in analgesia after lumbar medial branch block #1 (measured by numeric pain rating scale) after infusing saline
Change in low back pain score after Lumbar Medial Branch Block #2 | Approximately 2 weeks after Lumbar Medial Branch Block #1, and before Lumbar Medial Branch Radiofrequency Neurotomy
  Change in Numeric Pain Rating Scale score for low back pain after Lumbar Medial Branch Block #2
Change in low back pain score after Lumbar Medial Branch Radiofrequency Neurotomy | Baseline, then 6 weeks, 3 months, 6 months after Lumbar Medial Branch Radiofrequency Neurotomy
  Change in Numeric Pain Rating Scale score for low back pain after Lumbar Medial Branch Neurotomy
Change in McGill Pain Questionnaire-2 after Lumbar Medial Branch Radiofrequency Neurotomy | Baseline, then 6 weeks, 3 months, 6 months after Lumbar Medial Branch Radiofrequency Neurotomy
  Change in McGill Pain Questionnaire-2 score after Lumbar Medial Branch Radiofrequency Neurotomy
Change in MQS-III after Lumbar Medial Branch Radiofrequency Neurotomy | Baseline, then 6 weeks, 3 months, 6 months after Lumbar Medial Branch Radiofrequency Neurotomy
  Change in MQS-III score after Lumbar Medial Branch Radiofrequency Neurotomy
Change in Patient-Reported Outcomes Measurement Information System-29 after Lumbar Medial Branch Radiofrequency Neurotomy | Baseline, then 6 weeks, 3 months, 6 months after Lumbar Medial Branch Radiofrequency Neurotomy
  Change in Patient-Reported Outcomes Measurement Information System-29 score after Lumbar Medial Branch Radiofrequency Neurotomy

OTHER OUTCOMES:
Fluoroscopy evaluation for procedural integrity - Lumbar Medial Branch Block | during Lumbar Medial Branch Block procedure
  Fluoroscopic images of Lumbar Medial Branch Blocks will be collected to document procedural integrity.
  This measure is a binary (yes,no) describing whether the tip of the procedure needle is in contact with the anatomical target on each of the procedural images.
Fluoroscopy evaluation for procedural integrity, distance - Lumbar Medial Branch Radiofrequency Neurotomy | during Lumbar Medial Branch Radiofrequency Neurotomy procedure
  Fluoroscopic images of Lumbar Medial Branch Radiofrequency Neurotomy will be collected to document procedural integrity.
  This measure is the number of radiofrequency cannula widths between the anatomical target and the radiofrequency cannula.
Fluoroscopy evaluation for procedural integrity, displacement - Lumbar Medial Branch Radiofrequency Neurotomy | during Lumbar Medial Branch Radiofrequency Neurotomy procedure
  Fluoroscopic images of Lumbar Medial Branch Radiofrequency Neurotomy will be collected to document procedural integrity.
  This specific measure is the (x,y) coordinates of the proximal and distal ends of the radiofrequency cannula tip minus the (x,y) coordinates of the proximal and distal bounds of the target structure.

CONTACTS AND LOCATIONS:
Overall Officials: William E Rivers, DO, Principal Investigator — Tennessee Valley Healthcare System VA
Locations (1):
- VA Tennessee Valley Healthcare System, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data will only be accessed and analyzed by primary research team.

REFERENCES:
- [Background] Benedetti F. The opposite effects of the opiate antagonist naloxone and the cholecystokinin antagonist proglumide on placebo analgesia. Pain. 1996 Mar;64(3):535-543. doi: 10.1016/0304-3959(95)00179-4. PMID 8783319
- [Background] Cohen SP, Williams KA, Kurihara C, Nguyen C, Shields C, Kim P, Griffith SR, Larkin TM, Crooks M, Williams N, Morlando B, Strassels SA. Multicenter, randomized, comparative cost-effectiveness study comparing 0, 1, and 2 diagnostic medial branch (facet joint nerve) block treatment paradigms before lumbar facet radiofrequency denervation. Anesthesiology. 2010 Aug;113(2):395-405. doi: 10.1097/ALN.0b013e3181e33ae5. PMID 20613471
- [Background] Cohen SP, Stojanovic MP, Crooks M, Kim P, Schmidt RK, Shields CH, Croll S, Hurley RW. Lumbar zygapophysial (facet) joint radiofrequency denervation success as a function of pain relief during diagnostic medial branch blocks: a multicenter analysis. Spine J. 2008 May-Jun;8(3):498-504. doi: 10.1016/j.spinee.2007.04.022. Epub 2007 Jun 18. PMID 17662665
- [Background] Manchukonda R, Manchikanti KN, Cash KA, Pampati V, Manchikanti L. Facet joint pain in chronic spinal pain: an evaluation of prevalence and false-positive rate of diagnostic blocks. J Spinal Disord Tech. 2007 Oct;20(7):539-45. doi: 10.1097/BSD.0b013e3180577812. PMID 17912133
- [Background] Cohen SP, Doshi TL, Constantinescu OC, Zhao Z, Kurihara C, Larkin TM, Griffith SR, Jacobs MB, Kroski WJ, Dawson TC, Fowler IM, White RL, Verdun AJ, Jamison DE, Anderson-White M, Shank SE, Pasquina PF. Effectiveness of Lumbar Facet Joint Blocks and Predictive Value before Radiofrequency Denervation: The Facet Treatment Study (FACTS), a Randomized, Controlled Clinical Trial. Anesthesiology. 2018 Sep;129(3):517-535. doi: 10.1097/ALN.0000000000002274. PMID 29847426
- [Background] Boswell MV, Manchikanti L, Kaye AD, Bakshi S, Gharibo CG, Gupta S, Jha SS, Nampiaparampil DE, Simopoulos TT, Hirsch JA. A Best-Evidence Systematic Appraisal of the Diagnostic Accuracy and Utility of Facet (Zygapophysial) Joint Injections in Chronic Spinal Pain. Pain Physician. 2015 Jul-Aug;18(4):E497-533. PMID 26218947
- [Background] Kaptchuk TJ, Goldman P, Stone DA, Stason WB. Do medical devices have enhanced placebo effects? J Clin Epidemiol. 2000 Aug;53(8):786-92. doi: 10.1016/s0895-4356(00)00206-7. PMID 10942860
- [Background] Finniss D, Nicholas M, Brooker C, Cousins M, Benedetti F. Magnitude, response, and psychological determinants of placebo effects in chronic low-back pain: a randomised, double-blinded, controlled trial. Pain Rep. 2019 Jun 7;4(3):e744. doi: 10.1097/PR9.0000000000000744. eCollection 2019 May-Jun. PMID 31583358
- [Background] Zubieta JK, Bueller JA, Jackson LR, Scott DJ, Xu Y, Koeppe RA, Nichols TE, Stohler CS. Placebo effects mediated by endogenous opioid activity on mu-opioid receptors. J Neurosci. 2005 Aug 24;25(34):7754-62. doi: 10.1523/JNEUROSCI.0439-05.2005. PMID 16120776
- [Background] Bagley EE, Ingram SL. Endogenous opioid peptides in the descending pain modulatory circuit. Neuropharmacology. 2020 Aug 15;173:108131. doi: 10.1016/j.neuropharm.2020.108131. Epub 2020 May 15. PMID 32422213
- [Background] Petrovic P, Pleger B, Seymour B, Kloppel S, De Martino B, Critchley H, Dolan RJ. Blocking central opiate function modulates hedonic impact and anterior cingulate response to rewards and losses. J Neurosci. 2008 Oct 15;28(42):10509-16. doi: 10.1523/JNEUROSCI.2807-08.2008. PMID 18923027
- [Background] Colloca L. Placebo effects in pain. Int Rev Neurobiol. 2020;153:167-185. doi: 10.1016/bs.irn.2020.04.001. Epub 2020 Jun 9. PMID 32563287
- [Background] Bruehl S, Burns JW, Morgan A, Koltyn K, Gupta R, Buvanendran A, Edwards D, Chont M, Kingsley PJ, Marnett L, Stone A, Patel S. The association between endogenous opioid function and morphine responsiveness: a moderating role for endocannabinoids. Pain. 2019 Mar;160(3):676-687. doi: 10.1097/j.pain.0000000000001447. PMID 30562268
- [Background] Bruehl S, Burns JW, Koltyn K, Gupta R, Buvanendran A, Edwards D, Chont M, Wu YH, Qu'd D, Stone A. Are endogenous opioid mechanisms involved in the effects of aerobic exercise training on chronic low back pain? A randomized controlled trial. Pain. 2020 Dec;161(12):2887-2897. doi: 10.1097/j.pain.0000000000001969. PMID 32569082
- [Background] Wager TD, Scott DJ, Zubieta JK. Placebo effects on human mu-opioid activity during pain. Proc Natl Acad Sci U S A. 2007 Jun 26;104(26):11056-61. doi: 10.1073/pnas.0702413104. Epub 2007 Jun 19. PMID 17578917
- [Background] Wartolowska KA, Gerry S, Feakins BG, Collins GS, Cook J, Judge A, Carr AJ. A meta-analysis of temporal changes of response in the placebo arm of surgical randomized controlled trials: an update. Trials. 2017 Jul 12;18(1):323. doi: 10.1186/s13063-017-2070-9. PMID 28701195
- [Background] Kaplan M, Dreyfuss P, Halbrook B, Bogduk N. The ability of lumbar medial branch blocks to anesthetize the zygapophysial joint. A physiologic challenge. Spine (Phila Pa 1976). 1998 Sep 1;23(17):1847-52. doi: 10.1097/00007632-199809010-00008. PMID 9762741
- [Background] Dreyfuss P, Halbrook B, Pauza K, Joshi A, McLarty J, Bogduk N. Efficacy and validity of radiofrequency neurotomy for chronic lumbar zygapophysial joint pain. Spine (Phila Pa 1976). 2000 May 15;25(10):1270-7. doi: 10.1097/00007632-200005150-00012. PMID 10806505
- [Background] Dreyfuss P, Schwarzer AC, Lau P, Bogduk N. Specificity of lumbar medial branch and L5 dorsal ramus blocks. A computed tomography study. Spine (Phila Pa 1976). 1997 Apr 15;22(8):895-902. doi: 10.1097/00007632-199704150-00013. PMID 9127924
- [Background] McCormick ZL, Marshall B, Walker J, McCarthy R, Walega DR. Long-Term Function, Pain and Medication Use Outcomes of Radiofrequency Ablation for Lumbar Facet Syndrome. Int J Anesth Anesth. 2015;2(2):028. doi: 10.23937/2377-4630/2/2/1028. PMID 26005713
- [Background] MacVicar J, Borowczyk JM, MacVicar AM, Loughnan BM, Bogduk N. Lumbar medial branch radiofrequency neurotomy in New Zealand. Pain Med. 2013 May;14(5):639-45. doi: 10.1111/pme.12000. Epub 2012 Dec 28. PMID 23279154